CLINICAL TRIAL: NCT06931821
Title: Functional ElectroAnatomiC Isochronal Late Activation Mapping for Empiric VT Ablation Trial
Acronym: FACILE-VT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Roderick Tung, Chief, Division of Cardiology, and Director, Cardiovascular Clinical Research,, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003834
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sustained Monomorphic VT (MMVT); Recurrent Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Isochronal Late Activation Mapping; high-density mapping; deceleration zone
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial with 1:1 randomization to two strategies for ventricular tachycardia (VT) mapping and ablation.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High Density Voltage Mapping (Active Comparator): high-density voltage mapping will serve as the method to display the electroanatomic substrate for extensive and diffuse ablation within the low voltage area (<1.5 mV)
  Interventions: Device: High Density Voltage Mapping
- Isochronal Late Activation Mapping (ILAM) (Experimental): an isochronal late activation mapping (ILAM) display with automated last deflection annotation (EnSite X™) will be used to identify regions of isochronal crowding around a line of conduction block for targeted ablation therapy using a standard irrigated tip catheter (Flexability SE & Tactiflex catheters).
  Interventions: Device: Isochronal Late Activation Mapping (ILAM)

INTERVENTIONS:
Device: Isochronal Late Activation Mapping (ILAM) — an isochronal late activation mapping (ILAM) display with automated last deflection annotation (EnSite X™) will be used to identify regions of isochronal crowding around a line of conduction block for targeted ablation therapy using a standard irrigated tip catheter (Flexability SE & Tactiflex catheters)
  Arms: Isochronal Late Activation Mapping (ILAM)
Device: High Density Voltage Mapping — high-density voltage mapping will serve as the method to display the electroanatomic substrate for extensive and diffuse ablation within the low voltage area (<1.5 mV).
  Arms: High Density Voltage Mapping

SUMMARY:
This is a multicenter, prospective, parallel, randomized controlled trial to test for non-inferiority with an ILAM-guided VT ablation compared to conventional voltage- based ablation. The study has two treatment arms: conventional voltage mapping and ablation (control arm). In the investigational arm, the ablation strategy is guided by ILAM to target deceleration zones, blinded to voltage mapping. In the control arm, ablation will be performed to extensively ablate all low voltage regions (<1.5mV) during sinus rhythm, right ventricular (RV) pacing, or left ventricular (LV) pacing, with discretionary use of pacemapping and activation mapping. In both arms, mapping with be performed with a multielectrode catheter (HD Grid) and ablation will be performed using an irrigated tip catheter (FlexAbility SE or Tactiflex catheters).

In the control armonly voltage mapping displays will be utilized (blinded to functional ILAM and fractionation). High density mapping with automated last deflection annotation (Ensite X) will be performed in all patients randomized to ILAM approach during either sinus rhythm or RV pacing.

ELIGIBILITY:
Criteria

To participate in this clinical investigation, the subjects must meet all of the following inclusion criteria:

1. Patient is ≥18 years of age.
2. Able and willing to comply with all study requirements.
3. At least one documented episode of sustained MMVT (>30 sec) by either EGM or ECG (including Holter, or loop recorder) in the 6 months prior to enrollment.
4. Informed of the nature of the study, agreed to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical study site.
5. Refractory (i.e., not effective, not tolerated, or not desired) to at least one anti-arrhythmic medication (including, but not limited to beta blocker, mexiletine, amiodarone or sotalol) for treatment of MMVT.
6. Structural heart disease (ischemic or non-ischemic) with one of the following (a, b or c):

   1. Evidence of myocardial scar by echocardiography (segmental wall motion or wall thinning), CT (wall thinning) and/or MRI (presence of delayed enhancement /late gadolinium enhancement) . CT or MRI with scar is mandatory for inclusion of NICM., or
   2. Left ventricular ejection fraction (EF) <50% [documented within the last 6 months via transthoracic echocardiogram (TTE), MRI] with presence of scar, or
   3. Arrhythmogenic RV cardiomyopathy/dysplasia (per 2010 ARVC/D Task Force Criteria)

Exclusion Criteria

Subjects who meet any of the following exclusion criteria must be excluded from the clinical investigation:

1. Active infection (positive blood culture).
2. Patient is pregnant or nursing.
3. Cardiac surgery via sternotomy (CABG or valve repair/replacement) within 30 days prior to enrollment.
4. Contraindication to systemic anticoagulation (i.e., heparin, warfarin, or a direct thrombin inhibitor).
5. Currently receiving support via extracorporeal membrane oxygenation (ECMO) or ventricular assist device (VAD).
6. Left Ventriclar ejection fraction < 15%.
7. Stroke within 30 days or presence of LV thrombus within 1 month prior to enrollment.
8. Idiopathic VT or preprocedural imaging without scar (MRI or CT).
9. Limited life expectancy of 1 year or less.
10. Presence of mitral and aortic valves both mechanical.
11. Ventricular tachycardia secondary to electrolyte imbalance or any other reversible or non-cardiac cause.
12. Severe aortic stenosis or flail mitral valve with severed mitral regurgitation.
13. Thrombocytopenia (defined as platelet count <50,000/μl ) or coagulopathy.
14. Ventricular arrhythmias secondary to underlying channelopathies (LQTS, Brugada Syndrome).
15. Enrolled in an investigational study evaluating another device or drug that would confound the results of this study.
16. Other anatomic or co-morbid conditions that, in the investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow up requirement of 1 year, or impact the scientific integrity of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Inducibility for VT | after initial 25 minutes of ablation (minutes of radiofrequency)
  Inducibility for VT after initial 25 minutes of ablation (minutes of radiofrequency)
Recurrent VT | 1 year post procedure
  recurrent VT at 1 year
CV Hospitalization | 1 year post procedure
  Hospitalization due to Cardiovascular complications related to heart failure or arrhythmia at 1 year
Mortality | 1 year post procedure
  Mortality at 1 year
Procedure Related Safety | Duration of Hospitalization (up to 7 days)
  hematoma requiring transfusion, cardiac perforation, stroke, hemorrhage, pericardial effusion

SECONDARY OUTCOMES:
Individual assessment of four endpoints comprising the primary endpoint. | 1 year post procedure
  Individual assessment of four individual endpoints comprising the primary endpoint.
Total radiofrequency time delivered and procedural time. | Duration of Procedure
Reduction in VT burden | 1 year post procedure
Quality of Life improvement | 1 year post procedure
  The overall quality of life will be assessed using the SF-36 instrument, which includes 36 items rated on a 4-point Likert scale. In all nine subscales, lower scores indicate poorer outcomes in various areas, including physical functioning, social limitations due to physical or mental health issues, challenges related to work or daily activities, and feelings of nervousness, depression, fatigue, exhaustion, and pain.
Procedural complications | Duration of Hospitalization (up to 7 days)
  tamponade, hematoma requiring transfusion, stroke, emergent surgery
Length of stay in hospital from index procedure | Duration of Hospitalization (up to 7 days)
Rate of Acute Kidney Injury | 1 day post procedure
  Number of Participants with acute kidney injury, verified by creatinine checked the day after ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Tung, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL. 2013 ACCF/AHA guideline for the management of heart failure: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):1810-52. doi: 10.1161/CIR.0b013e31829e8807. Epub 2013 Jun 5. No abstract available. PMID 23741057
- [Background] Seiler J, Roberts-Thomson KC, Raymond JM, Vest J, Delacretaz E, Stevenson WG. Steam pops during irrigated radiofrequency ablation: feasibility of impedance monitoring for prevention. Heart Rhythm. 2008 Oct;5(10):1411-6. doi: 10.1016/j.hrthm.2008.07.011. Epub 2008 Jul 10. PMID 18929327
- [Background] Jais P, Maury P, Khairy P, Sacher F, Nault I, Komatsu Y, Hocini M, Forclaz A, Jadidi AS, Weerasooryia R, Shah A, Derval N, Cochet H, Knecht S, Miyazaki S, Linton N, Rivard L, Wright M, Wilton SB, Scherr D, Pascale P, Roten L, Pederson M, Bordachar P, Laurent F, Kim SJ, Ritter P, Clementy J, Haissaguerre M. Elimination of local abnormal ventricular activities: a new end point for substrate modification in patients with scar-related ventricular tachycardia. Circulation. 2012 May 8;125(18):2184-96. doi: 10.1161/CIRCULATIONAHA.111.043216. Epub 2012 Apr 4. PMID 22492578
- [Background] Jiang R, Beaser AD, Aziz Z, Upadhyay GA, Nayak HM, Tung R. High-Density Grid Catheter for Detailed Mapping of Sinus Rhythm and Scar-Related Ventricular Tachycardia: Comparison With a Linear Duodecapolar Catheter. JACC Clin Electrophysiol. 2020 Mar;6(3):311-323. doi: 10.1016/j.jacep.2019.11.007. Epub 2020 Jan 29. PMID 32192682
- [Background] Raiman M, Tung R. Automated isochronal late activation mapping to identify deceleration zones: Rationale and methodology of a practical electroanatomic mapping approach for ventricular tachycardia ablation. Comput Biol Med. 2018 Nov 1;102:336-340. doi: 10.1016/j.compbiomed.2018.07.012. Epub 2018 Jul 18. PMID 30033360
- [Background] Marcus FI, McKenna WJ, Sherrill D, Basso C, Bauce B, Bluemke DA, Calkins H, Corrado D, Cox MG, Daubert JP, Fontaine G, Gear K, Hauer R, Nava A, Picard MH, Protonotarios N, Saffitz JE, Sanborn DM, Steinberg JS, Tandri H, Thiene G, Towbin JA, Tsatsopoulou A, Wichter T, Zareba W. Diagnosis of arrhythmogenic right ventricular cardiomyopathy/dysplasia: proposed modification of the task force criteria. Circulation. 2010 Apr 6;121(13):1533-41. doi: 10.1161/CIRCULATIONAHA.108.840827. Epub 2010 Feb 19. PMID 20172911
- [Background] Irie T, Yu R, Bradfield JS, Vaseghi M, Buch EF, Ajijola O, Macias C, Fujimura O, Mandapati R, Boyle NG, Shivkumar K, Tung R. Relationship between sinus rhythm late activation zones and critical sites for scar-related ventricular tachycardia: systematic analysis of isochronal late activation mapping. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):390-9. doi: 10.1161/CIRCEP.114.002637. Epub 2015 Mar 4. PMID 25740836
- [Background] Tung R, Josephson ME, Bradfield JS, Shivkumar K. Directional Influences of Ventricular Activation on Myocardial Scar Characterization: Voltage Mapping With Multiple Wavefronts During Ventricular Tachycardia Ablation. Circ Arrhythm Electrophysiol. 2016 Aug;9(8):e004155. doi: 10.1161/CIRCEP.116.004155. PMID 27516464
- [Background] Tung R, Kim S, Yagishita D, Vaseghi M, Ennis DB, Ouadah S, Ajijola OA, Bradfield JS, Mahapatra S, Finn P, Shivkumar K. Scar voltage threshold determination using ex vivo magnetic resonance imaging integration in a porcine infarct model: Influence of interelectrode distances and three-dimensional spatial effects of scar. Heart Rhythm. 2016 Oct;13(10):1993-2002. doi: 10.1016/j.hrthm.2016.07.003. Epub 2016 Jul 5. PMID 27392944
- [Background] Nakahara S, Tung R, Ramirez RJ, Michowitz Y, Vaseghi M, Buch E, Gima J, Wiener I, Mahajan A, Boyle NG, Shivkumar K. Characterization of the arrhythmogenic substrate in ischemic and nonischemic cardiomyopathy implications for catheter ablation of hemodynamically unstable ventricular tachycardia. J Am Coll Cardiol. 2010 May 25;55(21):2355-65. doi: 10.1016/j.jacc.2010.01.041. PMID 20488307
- [Background] Tung R, Nakahara S, Ramirez R, Gui D, Magyar C, Lai C, Fishbein M, Shivkumar K. Accuracy of combined endocardial and epicardial electroanatomic mapping of a reperfused porcine infarct model: a comparison of electrofield and magnetic systems with histopathologic correlation. Heart Rhythm. 2011 Mar;8(3):439-47. doi: 10.1016/j.hrthm.2010.10.044. Epub 2010 Nov 4. PMID 21056123
- [Background] Tung R, Nakahara S, Maccabelli G, Buch E, Wiener I, Boyle NG, Carbucicchio C, Bella PD, Shivkumar K. Ultra high-density multipolar mapping with double ventricular access: a novel technique for ablation of ventricular tachycardia. J Cardiovasc Electrophysiol. 2011 Jan;22(1):49-56. doi: 10.1111/j.1540-8167.2010.01859.x. PMID 20653813
- [Background] Tung R, Vaseghi M, Frankel DS, Vergara P, Di Biase L, Nagashima K, Yu R, Vangala S, Tseng CH, Choi EK, Khurshid S, Patel M, Mathuria N, Nakahara S, Tzou WS, Sauer WH, Vakil K, Tedrow U, Burkhardt JD, Tholakanahalli VN, Saliaris A, Dickfeld T, Weiss JP, Bunch TJ, Reddy M, Kanmanthareddy A, Callans DJ, Lakkireddy D, Natale A, Marchlinski F, Stevenson WG, Della Bella P, Shivkumar K. Freedom from recurrent ventricular tachycardia after catheter ablation is associated with improved survival in patients with structural heart disease: An International VT Ablation Center Collaborative Group study. Heart Rhythm. 2015 Sep;12(9):1997-2007. doi: 10.1016/j.hrthm.2015.05.036. Epub 2015 May 30. PMID 26031376
- [Background] Al-Khatib SM, Daubert JP, Anstrom KJ, Daoud EG, Gonzalez M, Saba S, Jackson KP, Reece T, Gu J, Pokorney SD, Granger CB, Hess PL, Mark DB, Stevenson WG. Catheter ablation for ventricular tachycardia in patients with an implantable cardioverter defibrillator (CALYPSO) pilot trial. J Cardiovasc Electrophysiol. 2015 Feb;26(2):151-7. doi: 10.1111/jce.12567. Epub 2014 Nov 30. PMID 25332150
- [Background] Reddy VY, Reynolds MR, Neuzil P, Richardson AW, Taborsky M, Jongnarangsin K, Kralovec S, Sediva L, Ruskin JN, Josephson ME. Prophylactic catheter ablation for the prevention of defibrillator therapy. N Engl J Med. 2007 Dec 27;357(26):2657-65. doi: 10.1056/NEJMoa065457. PMID 18160685
- [Background] Kuck KH, Schaumann A, Eckardt L, Willems S, Ventura R, Delacretaz E, Pitschner HF, Kautzner J, Schumacher B, Hansen PS; VTACH study group. Catheter ablation of stable ventricular tachycardia before defibrillator implantation in patients with coronary heart disease (VTACH): a multicentre randomised controlled trial. Lancet. 2010 Jan 2;375(9708):31-40. doi: 10.1016/S0140-6736(09)61755-4. PMID 20109864
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Calkins H, Epstein A, Packer D, Arria AM, Hummel J, Gilligan DM, Trusso J, Carlson M, Luceri R, Kopelman H, Wilber D, Wharton JM, Stevenson W. Catheter ablation of ventricular tachycardia in patients with structural heart disease using cooled radiofrequency energy: results of a prospective multicenter study. Cooled RF Multi Center Investigators Group. J Am Coll Cardiol. 2000 Jun;35(7):1905-14. doi: 10.1016/s0735-1097(00)00615-x. PMID 10841242
- [Background] Aliot EM, Stevenson WG, Almendral-Garrote JM, Bogun F, Calkins CH, Delacretaz E, Della Bella P, Hindricks G, Jais P, Josephson ME, Kautzner J, Kay GN, Kuck KH, Lerman BB, Marchlinski F, Reddy V, Schalij MJ, Schilling R, Soejima K, Wilber D; European Heart Rhythm Association (EHRA); Registered Branch of the European Society of Cardiology (ESC); Heart Rhythm Society (HRS); American College of Cardiology (ACC); American Heart Association (AHA). EHRA/HRS Expert Consensus on Catheter Ablation of Ventricular Arrhythmias: developed in a partnership with the European Heart Rhythm Association (EHRA), a Registered Branch of the European Society of Cardiology (ESC), and the Heart Rhythm Society (HRS); in collaboration with the American College of Cardiology (ACC) and the American Heart Association (AHA). Heart Rhythm. 2009 Jun;6(6):886-933. doi: 10.1016/j.hrthm.2009.04.030. No abstract available. PMID 19467519
- [Background] Natale A, Raviele A, Al-Ahmad A, Alfieri O, Aliot E, Almendral J, Breithardt G, Brugada J, Calkins H, Callans D, Cappato R, Camm JA, Della Bella P, Guiraudon GM, Haissaguerre M, Hindricks G, Ho SY, Kuck KH, Marchlinski F, Packer DL, Prystowsky EN, Reddy VY, Ruskin JN, Scanavacca M, Shivkumar K, Soejima K, Stevenson WJ, Themistoclakis S, Verma A, Wilber D; Venice Chart members. Venice Chart International Consensus document on ventricular tachycardia/ventricular fibrillation ablation. J Cardiovasc Electrophysiol. 2010 Mar;21(3):339-79. doi: 10.1111/j.1540-8167.2009.01686.x. Epub 2010 Jan 15. No abstract available. PMID 20082650
- [Background] Xie J, Weil MH, Sun S, Tang W, Sato Y, Jin X, Bisera J. High-energy defibrillation increases the severity of postresuscitation myocardial dysfunction. Circulation. 1997 Jul 15;96(2):683-8. doi: 10.1161/01.cir.96.2.683. PMID 9244243
- [Background] Epstein AE, Kay GN, Plumb VJ, Dailey SM, Anderson PG. Gross and microscopic pathological changes associated with nonthoracotomy implantable defibrillator leads. Circulation. 1998 Oct 13;98(15):1517-24. doi: 10.1161/01.cir.98.15.1517. PMID 9769305
- [Background] Vergara P, Trevisi N, Ricco A, Petracca F, Baratto F, Cireddu M, Bisceglia C, Maccabelli G, Della Bella P. Late potentials abolition as an additional technique for reduction of arrhythmia recurrence in scar related ventricular tachycardia ablation. J Cardiovasc Electrophysiol. 2012 Jun;23(6):621-7. doi: 10.1111/j.1540-8167.2011.02246.x. Epub 2012 Apr 4. PMID 22486970
- [Background] Bilge AK, Ozben B, Demircan S, Cinar M, Yilmaz E, Adalet K. Depression and anxiety status of patients with implantable cardioverter defibrillator and precipitating factors. Pacing Clin Electrophysiol. 2006 Jun;29(6):619-26. doi: 10.1111/j.1540-8159.2006.00409.x. PMID 16784428
- [Background] Kamphuis HC, de Leeuw JR, Derksen R, Hauer RN, Winnubst JA. Implantable cardioverter defibrillator recipients: quality of life in recipients with and without ICD shock delivery: a prospective study. Europace. 2003 Oct;5(4):381-9. doi: 10.1016/s1099-5129(03)00078-3. PMID 14753636
- [Background] Sears SE Jr, Conti JB. Understanding implantable cardioverter defibrillator shocks and storms: medical and psychosocial considerations for research and clinical care. Clin Cardiol. 2003 Mar;26(3):107-11. doi: 10.1002/clc.4960260303. PMID 12685615
- [Background] Pacifico A, Hohnloser SH, Williams JH, Tao B, Saksena S, Henry PD, Prystowsky EN. Prevention of implantable-defibrillator shocks by treatment with sotalol. d,l-Sotalol Implantable Cardioverter-Defibrillator Study Group. N Engl J Med. 1999 Jun 17;340(24):1855-62. doi: 10.1056/NEJM199906173402402. PMID 10369848
- [Background] Connolly SJ, Dorian P, Roberts RS, Gent M, Bailin S, Fain ES, Thorpe K, Champagne J, Talajic M, Coutu B, Gronefeld GC, Hohnloser SH; Optimal Pharmacological Therapy in Cardioverter Defibrillator Patients (OPTIC) Investigators. Comparison of beta-blockers, amiodarone plus beta-blockers, or sotalol for prevention of shocks from implantable cardioverter defibrillators: the OPTIC Study: a randomized trial. JAMA. 2006 Jan 11;295(2):165-71. doi: 10.1001/jama.295.2.165. PMID 16403928